CLINICAL TRIAL: NCT07273825
Title: The Effect of Geranium Essential Oil Aromatherapy on Fatigue and Sleep Quality in Patients Undergoing Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Muhammadiyah Surakarta (Other)
Responsible Party: Principal Investigator, Fahrun Nur Rosyid, Head of Quality Assurance Group, Universitas Muhammadiyah Surakarta
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UMuhammadiyahSurakarta
Record Dates: First submitted 2025-11-20; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Aromatherapy (Geranium Essential Oil); Chronic Kidney Disease on Hemodialysis; End Stage Renal Disease (ESRD); Fatigue; Poor Sleep Quality; Aromatherapy
Keywords: Aromatherapy; Geranium Essential Oil; Fatigue; Hemodialysis; Sleep Quality
MeSH Terms: conditions — Kidney Failure, Chronic; Fatigue; Sleep Initiation and Maintenance Disorders | interventions — Aromatherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Placebo Comparator): Participants in this arm will receive placebo aromatherapy (odorless substance) during hemodialysis sessions. The placebo is administered in the same manner as the geranium essential oil aromatherapy to maintain consistency of procedures. No active essential oil components are present. Fatigue will be measured using the FACIT-F scale, and sleep quality will be evaluated using the Pittsburgh Sleep Quality Index (PSQI). After completing this phase, participants will cross over to the intervention arm according to the randomized sequence.
  Interventions: Other: Placebo Aromatherapy (Non-Geranium Neutral Oil)
- Geranium Essential Oil Aromatherapy Arm (Experimental): Participants in this arm will receive geranium essential oil aromatherapy during hemodialysis sessions. The aromatherapy is administered through inhalation of geranium essential oil during the treatment period. Fatigue will be assessed using the FACIT-F scale and sleep quality will be measured using the PSQI before and after the intervention. After the intervention phase, participants will cross over to the control arm according to the randomized schedule.
  Interventions: Other: Geranium Aromatherapy

INTERVENTIONS:
Other: Placebo Aromatherapy (Non-Geranium Neutral Oil) — The placebo aromatherapy uses a non-active neutral oil without geranium's aromatic compounds or therapeutic properties. The placebo oil has a mild scent designed to mimic the inhalation procedure without producing physiological effects. It is administered using the same method, duration, and frequency as the Geranium Essential Oil intervention to ensure blinding and maintain procedural consistency. This placebo serves as a comparison to evaluate the true effect of Geranium Essential Oil on fatigue and sleep quality in hemodialysis patients.
  Other Names: Neutral Aromatherapy Placebo
  Arms: Control Arm
Other: Geranium Aromatherapy — Geranium Essential Oil aromatherapy is administered through inhalation to provide relaxation effects aimed at reducing fatigue and improving sleep quality in patients undergoing hemodialysis. Geranium oil contains active components such as citronellol, geraniol, and linalool, which exhibit anti-inflammatory, analgesic, antioxidant, and calming properties. In this study, the intervention is applied before and/or during hemodialysis sessions using a randomized cross-over design to compare its effects on fatigue and sleep quality.
  Other Names: Geranium Essential Oil (GEO) Aromatherapy
  Arms: Geranium Essential Oil Aromatherapy Arm

SUMMARY:
Hemodialysis is a life-sustaining therapy for individuals with chronic kidney disease; however, it is often accompanied by adverse effects such as fatigue and poor sleep quality. Fatigue is one of the most frequently reported symptoms among hemodialysis patients and can significantly impair daily functioning, psychosocial wellbeing, and overall quality of life. Sleep disturbances are also common and may further exacerbate physical and emotional stress.

Aromatherapy using essential oils has been explored as a non-pharmacological intervention to reduce fatigue and improve sleep quality. Geranium essential oil contains active compounds such as geraniol, citronellol, and terpineol, which possess relaxing, anti-inflammatory, and analgesic properties. These characteristics indicate its potential to alleviate fatigue and promote better sleep.

This study aims to evaluate the effect of geranium essential oil aromatherapy on fatigue and sleep quality in patients undergoing hemodialysis. The study employs a randomized cross-over design involving 90 participants who meet predetermined inclusion criteria. Fatigue will be assessed using the Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F), and sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI). Assessments will be conducted before and after the intervention period.

The findings of this study are expected to provide scientific evidence supporting the use of geranium essential oil aromatherapy as a safe, accessible complementary therapy that may help reduce fatigue and improve sleep quality among hemodialysis patients.

DETAILED DESCRIPTION:
Chronic kidney disease continues to increase worldwide and represents a major contributor to global morbidity and mortality. Hemodialysis is a primary treatment modality for replacing impaired renal function; however, the procedure is associated with various complications, including fatigue and sleep disturbances. Fatigue is one of the most prevalent symptoms among hemodialysis patients, with reported rates ranging from 60% to 97%. It can arise from multiple factors, including anemia, duration of hemodialysis, nutritional status, comorbidities, and uremic neuropathy. Persistent fatigue negatively impacts physical functioning, emotional wellbeing, social interaction, and overall quality of life.

Sleep disturbances are also frequently experienced by patients undergoing hemodialysis. Poor sleep quality may worsen fatigue, impair daytime functioning, and contribute to psychological distress. Given the complex and chronic nature of these symptoms, non-pharmacological interventions are increasingly explored to support symptom management.

Aromatherapy represents one complementary approach that has shown promising effects in managing fatigue and sleep problems. Geranium essential oil contains biologically active compounds-such as geraniol, citronellol, and other terpenoid alcohols-that exhibit relaxing, anti-inflammatory, and analgesic effects. When inhaled, aromatic molecules stimulate olfactory receptors, triggering neural signaling to the limbic system, which plays a key role in emotional regulation, stress response, hormonal balance, and sleep cycles. This mechanism suggests potential therapeutic value for reducing fatigue and improving sleep.

Previous studies have indicated that aromatherapy can benefit hemodialysis patients by reducing fatigue, anxiety, and sleep disturbances, though evidence specifically regarding geranium essential oil remains limited. Therefore, this study aims to generate robust clinical data on the effectiveness of geranium aromatherapy in this population.

A randomized cross-over design will be used, involving 90 hemodialysis patients recruited from multiple dialysis centers. All participants will serve as both control and intervention subjects at different phases of the study, minimizing variability across individuals. Fatigue will be measured using the Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F), which evaluates physical and mental exhaustion affecting daily life. Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI), assessing multiple components of sleep behavior. Data analysis will include paired t-test, independent t-test, and Chi-Square test with a significance level of p < 0.05.

This study aims to:

1. evaluate the effect of geranium essential oil aromatherapy on fatigue levels in hemodialysis patients;
2. assess the effect of the intervention on sleep quality;
3. provide scientific justification for the use of geranium essential oil as a complementary and integrative therapy in hemodialysis care.

Planned outputs include publication in a reputable international journal, development of a book chapter, intellectual property registration, community health education activities, and undergraduate research theses. The overall goal is to contribute meaningful evidence for safe and effective complementary therapies derived from natural Indonesian plant products to enhance the quality of life of patients undergoing hemodialysis

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* Have no visual or hearing impairments.
* Provide informed consent to participate.
* Have undergone hemodialysis (HD) for at least 3 months.
* Regularly receive HD at the study site.
* Undergo HD at least 2 times per week. 'Experience moderate to severe fatigue.

Exclusion Criteria:

* Presence of respiratory disease.
* History of allergy to perfumes or fragrance products.
* Olfactory impairment (difficulty smelling).
* Use of other therapies for fatigue during the intervention period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Fatigue Score (FACIT-F Fatigue Scale) | Baseline (pre-intervention) and after each intervention phase (up to 30 days).
  Fatigue will be assessed using the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) scale, consisting of 13 items rated on a 0-4 Likert scale. Total scores reflect fatigue severity, with lower scores indicating worse fatigue. Measurements will be taken before and after the intervention and placebo periods in the randomized cross-over design.

SECONDARY OUTCOMES:
Change in Sleep Quality Score (Pittsburgh Sleep Quality Index - PSQI) | Baseline (pre-intervention) and after each intervention phase (up to 30 days)
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), which evaluates subjective sleep quality, sleep latency, sleep duration, disturbances, use of sleep medication, and daytime dysfunction. Higher scores indicate poorer sleep quality. Assessments will be conducted before and after each intervention and placebo phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Universitas Muhammadiyah Surakarta, Sukoharjo, Centre Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains sensitive clinical information from hemodialysis patients and cannot be sufficiently de-identified to ensure participant privacy. Only aggregated results will be made available through publications.